CLINICAL TRIAL: NCT03953456
Title: A Double-Blind, Placebo-Controlled, Cross-over Phase II Study to Evaluate the Effect of a 6-week Elafibranor (120mg) Treatment Administered Once Daily on Hepatic Lipid Composition in Subjects With Nonalcoholic Fatty Liver (NAFL)
Brief Title: Study to Evaluate the Effect of Elafibranor on Hepatic Lipid Composition in Subjects With Nonalcoholic Fatty Liver (NAFL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Continuation of the trial cannot serve a scientific purpose
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GFT505-219-8; 2019-000645-12 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Non-Alcoholic Fatty Liver
Keywords: Hepatic lipid composition; Elafibranor; Hepatic Glucose Production
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over (placebo or elafibranor [GFT505]) placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigator, subject, and study personnel will be blinded to the treatment.
  Identification numbers will be assigned to a subject at the Screening Visit. Upon completion of the Screening Visits, eligible subjects will be randomly assigned to Sequence Group A or Group B, defining the order of treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elafibranor 120mg followed by placebo (Experimental): Participants will first receive elafibranor 120mg for 6 weeks. After a washout period of 4-6 weeks, they will then receive placebo for 6 weeks
  Interventions: Drug: elafibranor 120mg; Drug: Placebo
- placebo followed by elafibranor 120mg (Placebo Comparator): Participants will first receive placebo for 6 weeks. After a washout period of 4-6 weeks, they will then receive elafibranor 120mg for 6 weeks
  Interventions: Drug: elafibranor 120mg; Drug: Placebo

INTERVENTIONS:
Drug: elafibranor 120mg — elafibranor 120mg is a coated tablet for oral administration, once daily
  Other Names: GFT505
Drug: Placebo — Placebo is a coated tablet for oral administration, once daily

SUMMARY:
This randomized, double-blind, cross-over (placebo or elafibranor [GFT505]) placebo-controlled study, will evaluate the effect on hepatic lipid composition and safety of elafibranor 120 mg quaque die (QD) versus placebo in an adult NAFL population after 6 weeks of treatment with a 4-week wash-out period. This study will achieve mechanistic information about the mode of action of Elafibranor on the (lipid) metabolism in the human fatty liver

ELIGIBILITY:
Inclusion Criteria:

* Males or post-menopausal females aged from 40-75 years inclusive at first Screening Visit. (Post-menopausal defined as: subject should be surgically sterilized at least 6 months or no spontaneous menses for at least 1 year prior to screening)
* Must provide signed written informed consent and agrees to comply with the study protocol.
* Liver fat percentage ≥ 5 percent (as measured with Magnetic Resonance Spectroscopy)
* 25.0 ≤ BMI ≤ 38.0 kg/m^2
* Stable dietary habits and physical activity pattern (over 3 months prior to Screening Visit)
* Subject agrees not to change dietary habits and physical activity pattern, to follow diet and lifestyle recommendations and not to consume or use illicit drugs during the study up to end of treatment.

Exclusion Criteria:

Medical history:

* Documented weight loss of more than 5 percent during the 6-month period prior to Screening Visit
* Contra-indications for magnetic resonance imaging / spectroscopy
* Known history of Type 1 and 2 diabetes
* Known chronic heart failure (Grade I to IV of New York Heart Association classification)
* History of clinically significant acute cardiac event within 6 months prior to Screening Visit such as: stroke, transient ischemic attack, or coronary heart disease (angina pectoris, myocardial infarction, revascularization procedures)
* Uncontrolled hypertension despite optimal antihypertensive therapy
* Other well documented causes of chronic liver disease according to standard diagnostic procedures.
* Symptoms of clinical depression
* Other concurrent medical (e.g., immunological, neoplastic, endocrine, hematological, gastrointestinal or neurological) or psychiatric condition, which, in the opinion of the Investigator, would place the subject at increased risk, preclude obtaining voluntary consent/assent or compliance with required study procedures, or would confound the objectives of study
* Known hypersensitivity to the investigation product or any of its formulation excipients

Concomitant medications and lifestyle:

* Fibrates are not permitted from 8 weeks before Screening up to end of treatment. Subjects taking statins or ezetimibe prior to Screening Visit 1 may participate if the dose has been stable for 3 months prior to Screening Visit 1 and no dose adjustments are anticipated
* Currently taking drugs that can induce steatosis/steatohepatitis including, but not restricted to: corticosteroids (parenteral & oral chronic administration only), amiodarone (Cordarone), tamoxifen (Nolvadex), and methotrexate (Rheumatrex, Trexall), which are not permitted 30 days prior to Screening and up to end of treatment
* Subjects receiving thiazolidinediones (glitazones [pioglitazone, rosiglitazone])
* Currently taking any medication that could interfere with study medication absorption, distribution, metabolism, or excretion or could lead to induction or inhibition of microsomal enzymes, e.g., indomethacin, which are not permitted from Randomization until end of treatment
* Any medication use known to interfere with glucose homeostasis/metabolism
* Smoking
* Current or recent history (<5years) of significant alcohol consumption. For men, significant consumption is typically defined as higher than 30 g pure alcohol per day. For women, it is typically defined as higher than 20 g pure alcohol per day
* Subjects who have donated blood or blood products within the previous month prior to screening or who plan to donate blood or blood products at any time during the trial and in the month following the end of the study
* Is participating in any other study and have received any other investigational drug or device within 30 days prior to Screening or are taking part in a non-medication study which, in the opinion of the Investigator, would interfere with study compliance or outcome assessments
* Subjects who cannot be contacted in case of emergency

In addition to the above criteria, subject should not present any of the following biological exclusion criteria:

* Positive anti-human immunodeficiency virus (HIV) antibody
* Positive hepatitis B surface antigen
* Positive hepatitis C Virus (HCV) antibody
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >5 x upper limit of normal (ULN)
* Conjugated bilirubin > 1.50mg/dL due to altered hepatic function Note: Gilbert Disease subjects are allowed into the study
* International normalized ratio >1.40 due to altered hepatic function
* Platelet count <100,000/mm^3 due to portal hypertension
* Serum creatinine levels >1.53 mg/dL in males and >1.24 mg/dL in females
* Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as subjects with markers of kidney damage or estimated glomerular filtration rate (eGFR) of less than 60 ml/min/1.73 m^2)
* Unexplained serum creatine phosphokinase (CPK) >2 x ULN. In case of explained elevated CPK >2 x ULN, the measurement can be repeated prior to Randomization. In this case, retest should be performed within 1 to 2 weeks after initial test. A CPK retest >2 x ULN leads to exclusion
* Hemoglobin A1c (HbA1C) > 6.4% and/or fasting plasma glucose (FGP) > 126 mg/dl

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Change in relative amount of saturated fatty acids in the liver | After 6 weeks
  Relative amount of saturated fatty acids (SFA) in the liver measured by Magnetic Resonance Spectroscopy (1H-MRS) at the end of 6 weeks treatment period

SECONDARY OUTCOMES:
Change in hepatic insulin sensitivity | After 6 weeks
  Hepatic insulin sensitivity measured by Hepatic Glucose Production (HGP) at the end of 6 weeks treatment period
Glucose homeostasis markers | After 6 weeks
  Fasting glycemia
Glucose homeostasis markers | After 6 weeks
  HbA1c
Glucose homeostasis markers | After 6 weeks
  Fasting insulinemia
Glucose homeostasis markers | After 6 weeks
  C-peptide
Glucose homeostasis markers | After 6 weeks
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) index
Glucose homeostasis markers | After 6 weeks
  Fructosamine
Lipid metabolism markers | After 6 weeks
  Triglycerides (TG)
Lipid metabolism markers | After 6 weeks
  Total cholesterol (TC)
Lipid metabolism markers | After 6 weeks
  High density lipoprotein-cholesterol (HDL-C)
Lipid metabolism markers | After 6 weeks
  Low density lipoprotein-cholesterol (LDL-C)
Lipid metabolism markers | After 6 weeks
  Non-HDL-C
Lipid metabolism markers | After 6 weeks
  Free fatty acid (FFA)
Inflammatory markers | After 6 weeks
  High sensitivity C-reactive protein (hs-CRP)
Inflammatory markers | After 6 weeks
  Fibrinogen
Inflammatory markers | After 6 weeks
  Haptoglobin
Liver function | After 6 weeks
  Alanine aminotransferase (ALT)
Liver function | After 6 weeks
  Aspartate aminotransferase (AST)
Liver function | After 6 weeks
  Gamma glutamyl transferase (GGT)
Liver function | After 6 weeks
  Alkaline phosphatase (ALP)
Liver function | After 6 weeks
  Total and conjugated bilirubin
Renal function | After 6 weeks
  Creatinine
Renal function | After 6 weeks
  Estimated glomerular filtration rate (using Modification of Diet in Renal Disease (MDRD) formula)
Renal function | After 6 weeks
  Blood urea nitrogen
Renal function | After 6 weeks
  Albumin
Renal function | After 6 weeks
  Uric acid
Renal function | After 6 weeks
  Total proteins
Body weight | After 6 weeks
Body Mass Index | After 6 weeks
Waist circumference | After 6 weeks
Incidence and severity of treatment emergent adverse events (TEAEs) and their relationship to study drug | After 6 weeks
Incidence of clinically meaningful changes from baseline in safety laboratory parameters, and vital signs | After 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Birman, MD, Study Director — Genfit
Locations (1):
- NUTRIM School of Nutrition and Translational Research in Metabolism, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided